CLINICAL TRIAL: NCT04580719
Title: Women and Women's Hygienic Protection: Evaluation of Women's Practices, Knowledge and Expectations for Intimate Protection
Acronym: R-PO19076
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19076
Record Dates: First submitted 2019-07-18; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-06

CONDITIONS: Intimate Protections
Keywords: intimate protections; CHU REIMS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patiente: Patients aged 18 to 50, presenting menstrual cycles, consulting in the obstetrics and gynecology department of the University Hospital of Reims whatever the reason for consultation can participate in the study after signing the consent of no opposition. Participation in the study will not change the patient's medical management.

SUMMARY:
Intimate protections are designed to absorb menstrual flow during menstruation. A woman will use an average of 6,000 intimate protections during her lifetime. Intimate protections are classified into two categories: internal intimate protections including tampon, menstrual cup, menstrual sponge, and external intimate protections including disposable or washable sanitary pads, panty liner, menstrual panty. The choice and use of a type of intimate protection will depend on multiple factors specific to each woman. Due to a growing media interest in this area, women have become extremely critical and suspicious of these devices, particularly about the Toxic Shock Syndrome, attributed to the use of tampon in women previously colonized vaginally by strain of toxin-producing Staphylococcus aureus (Toxic shock syndrome toxin-1 (TSST-1)). Similarly, chemical residues have been found in sanitary napkins.

As a result, women's expectations have changed and there is a greater demand for transparency with regard to intimate protection of their composition and their potential health risks. Women want more and more alternative to conventional intimate protections in today's climate of increasing environmental awareness.

It is a cross-sectional, observational, prospective, unicentric inclusion study (CHU de Reims). The primary objective is to describe women's intimate protection practices. The secondary objectives are to study the determinants of women's choice for intimate protection, to describe women's knowledge of the potential risks of these intimate protections. and women's information sources on intimate protections. Finally describe the expectations of women in terms of intimate protections. The results are intended to give a photograph of the practices and knowledge of women consulting in the Obstetrics and Gynecology Department of the University Hospital of Reims concerning intimate protections.

Patients aged 18 to 50, presenting menstrual cycles, consulting in the obstetrics and gynecology department of the University Hospital of Reims whatever the reason for consultation can participate in the study after signing the consent of no opposition. Participation in the study will not change the patient's medical management. Participation in the study will result in the completion of a questionnaire concerning intimate protections. The filling time of the questionnaire is estimated at 10 minutes.

This subject is evolving with a growing awareness of women on the management of their rules, the products used, their potential risks and the environment. This study will allow us to see if women are really informed and feel concerned by these changes. And in the end, find out if they are ready to turn to intimate protections called "alternatives" The results will give us a vision of the expectations of our patients in this area as well as the information received, and thus allow us to publish an information guide and good practices of the intimate protections available in the waiting rooms of our consultations.

In addition, this study will allow health professionals to discuss this subject more easily and easily with their patients.

ELIGIBILITY:
inclusion criteria :

* aged 18 to 50
* presenting menstrual cycles

exclusion criteria :

- not signing the consent of no opposition

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18 to 50, presenting menstrual cycles, consulting in the obstetrics and gynecology department of the University Hospital of Reims whatever the reason for consultation can participate in the study after signing the consent of no opposition. Participation in the study will not change the patient's medical management.
Sampling Method: Non-Probability Sample
Enrollment: 1153 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Use of tampon | Day 0
  Number of patients using tampon as hygienic protection
Use of menstrual cup menstrual sponge | Day 0
  Number of patients using menstrual cup as hygienic protection
Use of menstrual sponge | Day 0
  Number of patients using menstrual sponge as hygienic protection
Use of disposable sanitary pads | Day 0
  Number of patients using disposable sanitary pads as hygienic protection
Use of washable sanitary pads | Day 0
  Number of patients using washable sanitary pads as hygienic protection
Use of panty liner | Day 0
  Number of patients using panty liner as hygienic protection
Use of menstrual panty | Day 0
  Number of patients using menstrual panty as hygienic protection

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France